CLINICAL TRIAL: NCT03073772
Title: Effects on Cognitive Function, Estimated as a Global Brain Score, by Cognitive and Physical Fitness Training Added to a Multimodal Rehabilitation Program for Patients With Exhaustion Disorder
Brief Title: Rehabilitation for Improved Cognition
Acronym: RECO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Västerbotten County Council, Sweden (Other Government); Swedish Social Insurance Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REHSAM 99368-2009/RS09
Record Dates: First submitted 2017-02-22; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-02

CONDITIONS: Exhaustion; Syndrome; Burnout Syndrome
MeSH Terms: conditions — Syndrome; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continued multimodal rehabilitation (No Intervention): No addition of extra training in this group. Only ordinary continued multimodal rehabilitation.
- Computer-based cognitive training (Active Comparator): This arm also consisted of continued multimodal rehabilitation.
  Interventions: Behavioral: Computer-based cognitive training
- Physical fitness training (Active Comparator): This arm also consisted of continued multimodal rehabilitation.
  Interventions: Behavioral: Physical fitness training

INTERVENTIONS:
Behavioral: Computer-based cognitive training — A total of 36 training sessions, approximately 20 minutes long each. Five different tasks were used in training all tapping different aspects of cognitive control such as updating, shifting, visuo-spatial working memory and episodic memory binding.
  Arms: Computer-based cognitive training
Behavioral: Physical fitness training — A total of 36 training sessions, approximately 40 minutes long each, with physical fitness training performed as group indoor cycling. The participants were instructed to attain a load of approximately 65-80% of their maximum heart rate.
  Arms: Physical fitness training

SUMMARY:
Many patients with exhaustion disorders continue to have significant difficulties with attention and memory function which reduce their work ability. This randomized study investigates whether the addition of a 12-week period of specific cognitive training or physical fitness training could further enhance cognitive function in patients with exhaustion disorder participating in a multimodal rehabilitation program.

DETAILED DESCRIPTION:
This study was performed at The Stress Rehabilitation Clinic at the University hospital of Umeå. In total 161 patients with diagnosed exhaustion disorder were recruited consecutively to the study from March 2010 until June 2013. Participants were all in age span 18-60 years old, had an ongoing employment and were assessed as suitable for a 24-week multimodal rehabilitation, which consisted of cognitive behavioural therapy in group (maximum eight persons), prescription of physical activity/exercise (FaR©) and vocational measures with rehabilitation meetings. A randomization by group was performed after 12 weeks of multimodal rehabilitation to one of three conditions; A/ continued multimodal rehabilitation, B/ addition of a computer-based cognitive training, and C/ addition of physical fitness training. The added training was performed during the last 12 weeks of rehabilitation (week 12 to 24) and with three weekly training occasions. Primary endpoint was change in cognitive functioning, estimated as a global brain score. Secondary endpoints were changes in different specific neuropsychological tasks, estimated psychological wellbeing, physical capacity, work ability, health-related quality of life and cost-effectiveness. A long-term follow-up was performed one year after termination of the interventions (at week 76).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed exhaustion disorder according to criteria established by the Swedish National Board of Health and Welfare
* 18 - 60 years of age
* Current employment
* Considered suitable for multimodal rehabilitation in group

Exclusion Criteria:

* Need of other treatment or rehabilitation
* Abuse of alcohol or drugs
* Participation in another intervention study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Short-term change in global brain score | Week 12 and 24
  The global brain score was calculated from ten neuropsychological tasks covering different domains in cognitive functioning
Long-term change in global brain score | Week 12, 24 and 76, mixed model with several time points used to estimate long-term effects
  The global brain score was calculated from ten neuropsychological tasks covering different domains in cognitive functioning

SECONDARY OUTCOMES:
Short-term change in "letter memory running span task" | Week 12 and 24
  A measure of the updating functioning
Long-term change in "letter memory running span task" | Week 12, 24 and 76, mixed model with several time points used to estimate long-term effects
  A measure of the updating functioning
Short-term change in "3-back task" | Week 12 and 24
  A measure of the updating functioning
Long-term change in "3-back task" | Week 12, 24 and 76, mixed model with several time points used to estimate long-term effects
  A measure of the updating functioning
Short-term change in the "colour word interference test (the Stroop test)" | Week 12 and 24
  A measure of the inhibition functioning, from D-KEFS
Long-term change in the "colour word interference test (the Stroop test)" | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  A measure of the inhibition functioning, from D-KEFS
Short-term change in the "trail making test" | Week 12 and 24
  A measure of attentional shifting, from D-KEFS
Long-term change in the "trail making test" | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  A measure of attentional shifting, from D-KEFS
Short-term change in the "digit span forward test" | Week 12 and 24
  A measure of the working memory, from WAIS-R
Long-term change in the "digit span forward test" | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  A measure of the working memory, from WAIS-R
Short-term change in the "digit span backward test" | Week 12 and 24
  A measure of the working memory, from WAIS-R
Long-term change in the "digit span backward test" | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  A measure of the working memory, from WAIS-R
Short-term change in the "letter-number sequencing" test | Week 12 and 24
  A measure of the working memory, from WAIS-III
Long-term change in the "letter-number sequencing" test | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  A measure of the working memory, from WAIS-III
Short-term change in the "recall of concrete nouns" test (Buschke's selective reminding procedure) | Week 12 and 24
  A measure of the episodic memory
Long-term change in the "recall of concrete nouns" test (Buschke's selective reminding procedure) | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  A measure of the episodic memory
Short-term change in the "digit symbol" test | Week 12 and 24
  A measure of perceptual speed, from WAIS-R
Long-term change in the "digit symbol" test | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  A measure of perceptual speed, from WAIS-R
Short-term change in "Raven's advanced progressive matrices" | Week 12 and 24
  A measure of non-verbal reasoning ability
Long-term change in "Raven's advanced progressive matrices" | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  A measure of non-verbal reasoning ability
Short-term change in Shirom Melamed Burnout Questionnaire | Week 12 and 24
  A burnout measure
Long-term change in Shirom Melamed Burnout Questionnaire | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  A burnout measure
Short-term change in Short Form 36 item Health Questionnaire | Week 12 and 24
  Health-related quality of life estimate
Long-term change in Short Form 36 item Health Questionnaire | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  Health-related quality of life estimate
Short-term change in Checklist Individual Strength Questionnaire | Week 12 and 24
  Measure of fatigue
Long-term change in Checklist Individual Strength Questionnaire | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  Measure of fatigue
Short-term change in Hospital Anxiety and Depression Scale, HAD-S | Week 12 and 24
  A measure of anxiety and depression
Long-term change in Hospital Anxiety and Depression Scale, HAD-S | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  A measure of anxiety and depression
Short-term change in aerobic capacity | Week 12 and 24
  A submaximal cycle ergometer test performed to estimate maximal oxygen uptake
Long-term change in aerobic capacity | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  A submaximal cycle ergometer test performed to estimate maximal oxygen uptake
Short-term change in work ability | Week 12 and 24
  Work Ability Index questionnaire, short version
Long-term change in work ability | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  Work Ability Index questionnaire, short version
Long-term total sick leave change | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  Information about sick leave from registers at the Social Insurance Agency in Sweden
Long-term cost-effectiveness | Week 12, 24 and 76, mixed model with several time points to estimate long-term effects
  Estimation of Changes in Quality Adjusted Life Years by using the Short Form-(36) Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Lisbeth Slunga Järvholm, MD, Ass Prof, Principal Investigator — Umeå University
Locations (1):
- Stress Rehabilitation Clinic, Umeå university hospital, Västerbotten county council, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nelson A, Aronsson I, Tillfors M, Neely AS, Gavelin HM. The experienced route to cognitive health: Cognitive recovery in persons with prior stress-related Exhaustion disorder. BMC Psychiatry. 2025 Apr 14;25(1):375. doi: 10.1186/s12888-025-06713-7. PMID 40229758
- [Derived] Nelson A, Gavelin HM, Boraxbekk CJ, Eskilsson T, Josefsson M, Slunga Jarvholm L, Neely AS. Subjective cognitive complaints in patients with stress-related exhaustion disorder: a cross sectional study. BMC Psychol. 2021 May 18;9(1):84. doi: 10.1186/s40359-021-00576-9. PMID 34006315
- [Derived] Malmberg Gavelin H, Eskilsson T, Boraxbekk CJ, Josefsson M, Stigsdotter Neely A, Slunga Jarvholm L. Rehabilitation for improved cognition in patients with stress-related exhaustion disorder: RECO - a randomized clinical trial. Stress. 2018 Jul;21(4):279-291. doi: 10.1080/10253890.2018.1461833. Epub 2018 Apr 25. PMID 29693483
- [Derived] Eskilsson T, Slunga Jarvholm L, Malmberg Gavelin H, Stigsdotter Neely A, Boraxbekk CJ. Aerobic training for improved memory in patients with stress-related exhaustion: a randomized controlled trial. BMC Psychiatry. 2017 Sep 2;17(1):322. doi: 10.1186/s12888-017-1457-1. PMID 28865430